CLINICAL TRIAL: NCT01663376
Title: Effects of Adipose Tissue Derived Stem Cells Implantation in Patients With Critical Limb Ischemia
Brief Title: Safety and Effect of Adipose Tissue Derived Mesenchymal Stem Cells Implantation in Patients With Critical Limb Ischemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: R-Bio (Industry)
Collaborators: Pusan National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSC-MSCs-CLI
Record Dates: First submitted 2012-08-08; First posted 2012-08-13 (Estimated); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Autologous Adipose Tissue derived MSCs Transplantation — Intramuscular injection of Autologous Adipose Derived Mesenchymal Stem Cells. Dose : 1x10e8 ~3x10e8 cells

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of autologous transplantation of Adipose Tissue derived Mesenchymal stem cells (MSCs) in patient with critical limb ischemia

ELIGIBILITY:
Inclusion Criteria:

* At least 6 months since the onset CLI(Chronic ASO or Buerger disease)
* Patients with luminal stenosis > 50% by leg angiography
* Age is between 20 and 80
* Patients whose Rutherford's class is II-4, III-5 or III-6 (Patients with rest pain or ischemic ulcer/necrosis)
* Patients for whom angioplasty and bypass surgery are not indicated because of anatomical or procedural reasons or frequent reocclusion/restenosis following traditional revascularization
* Patients who can give informed consent themselves in writing

Exclusion Criteria:

* Previous or current history of neoplasm or comorbidity that could impact the patient's survival
* Detection of proximal source of emboli including atrial fibrillation
* Primary hematologic disease, including hypercoagulable states
* Detection of proliferative retinopathy
* Entrapment syndrome
* Alcohol abuse, cocaine amphetamine etc.
* Detection of osteomyelitis
* Uncontrolled DM

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-01; Primary Completion 2010-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Major Adverse Events Analysis (MAEs) | 48 weeks
  To evaluate the change of treated critical limb ischemia before cell implantation and at 3, 6, 12 months post injection of MSCs

SECONDARY OUTCOMES:
Ankle-Brachial Index (ABI) | 48 weeks
  To evaluate the change of treated critical limb ischemia before cell implantation and at 3, 6, 12 months post injection of MSCs.
Digital subtraction angiography (DSA) | 48 weeks
  To evaluate the change of treated critical limb ischemia before cell implantation and at 3, 6, 12 months post injection of MSCs.
Thermography | 48 weeks
  To evaluate the change of treated critical limb ischemia before cell implantation and at 3, 6, 12 months post injection of MSCs.
Wong-Baker FACES Pain Rating Score | 48 weeks
  To evaluate the change of treated critical limb ischemia before cell implantation and at 3, 6, 12 months post injection of MSCs.
Treadmill test | 48 weeks
  To evaluate the change of treated critical limb ischemia before cell implantation and at 3, 6, 12 months post injection of MSCs.

CONTACTS AND LOCATIONS:
Overall Officials: Han Cheol Lee, M.D. & Ph.D., Principal Investigator — Pusan National University Hospital
Locations (1):
- Pusan National University Hospital, Pusan, South Korea

REFERENCES:
- [Result] Lee HC, An SG, Lee HW, Park JS, Cha KS, Hong TJ, Park JH, Lee SY, Kim SP, Kim YD, Chung SW, Bae YC, Shin YB, Kim JI, Jung JS. Safety and effect of adipose tissue-derived stem cell implantation in patients with critical limb ischemia: a pilot study. Circ J. 2012;76(7):1750-60. doi: 10.1253/circj.cj-11-1135. Epub 2012 Apr 12. PMID 22498564